CLINICAL TRIAL: NCT03047031
Title: An Active Surveillance to Monitor the Real World Safety in Indian Patients Prescribed Nintedanib for the Treatment of Idiopathic Pulmonary Fibrosis
Brief Title: Post Marketing Surveillance of Nintedanib in Indian Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0280
Record Dates: First submitted 2017-02-07; First posted 2017-02-08 (Estimated); Results first posted 2024-08-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib; pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- All nintedanib treated patients (group B + group C)
  Interventions: Drug: Nintedanib
- Group II- pirfenidone patients
  Interventions: Drug: Pirfenidone
- Group III - pirfenidone patients
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Nintedanib — Nintedanib
  Groups: All nintedanib treated patients (group B + group C)
Drug: Pirfenidone — Pirfenidone
  Groups: Group II- pirfenidone patients; Group III - pirfenidone patients

SUMMARY:
This is an active surveillance study to monitor the real world safety of nintedanib in Indian patients with Idiopathic Pulmonary Fibrosis. The safety of nintedanib has been assessed in clinical trials.This active surveillance aims to collect the safety data of 200 IPF patients treated with nintedanib in approved indication after the commercial availability of the drug in India (23rd January 2017). The objective is to look at safety of nintedanib in the real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented diagnosis of Idiopathic Pulmonary Fibrosis (IPF) based upon ATS/ERS/JRS/ALAT 2011 guidelines (nintedanib naïve or pirfenidone pre-treated) who have initiated or will initiate nintedanib according to the package insert after the commercial availability of drug in India (23rd January 2017).
* Patients in whom it is possible to obtain voluntary informed consent either from the patient or patient's legally authorised representative (applicable for Group B and C patients).
* Patients in whom data collection is possible from the medical records (applicable for Group A and B patients)
* Further inclusion criteria apply

Exclusion Criteria:

* Patients who were previously treated with nintedanib.
* Patients who have initiated or will initiate nintedanib concomitantly with pirfenidone..
* Patients who are participating in a clinical trial.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This active surveillance will include all IPF patients treated with nintedanib per the inclusion/exclusion criteria at selected centres during the first two years after the commercial availability of the drug.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- India (8):
  - Asthma Bhawan, Jaipur
  - National Allergy Asthma Bronchitis Institute, Kolkata, Kolkata
  - CK Birla Hospitals, The Calcutta Medical Research Institute, Kolkata
  - King George Medical University, Lucknow
  - Midland Healthcare and Research Centre, Lucknow
  - Bhatia Hospital, Mumbai
  - P.D. Hinduja National Hospital, Mumbai
  - Grant Medical Foundation, Ruby Hall Clinic, Pune

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This active surveillance study aimed to collect the safety data of Idiopathic Pulmonary Fibrosis (IPF) patients who were treated with nintedanib in approved indication after the commercial availability of the drug in India (23rd January 2017).
Pre-assignment Details: No patients were enrolled in Group A (nintedanib) & Group I (pirfenidone). The nintedanib patients in group B and group C were combined together in the participant flow and baseline characteristics, since the outcome measures and the adverse events were planned in the protocol of the study to be reported for all nintedanib treated patients.
Groups:
- All Nintedanib Treated Patients (Group B + Group C): This arm includes the patients who started treatment with nintedanib after 23rd January 2017 and were continuing the drug at the time of participation in the active surveillance (group B) and patients who were newly prescribed nintedanib at the time of participation in the active surveillance (group C). Initial dose in adult patients was Nintedanib 150 milligram (mg) twice daily orally administered with food in morning and evening. According to the Indian label the dosage could be reduced to nintedanib 100 mg twice daily according to the patient's symptoms or in case of adverse events.
- Group II- Pirfenidone Patients: This arm includes patients who started treatment with pirfenidone after the 23rd of January 2017 and are continuing the drug treatment at the time of participation in the active surveillance.
- Group III - Pirfenidone Patients: This arm includes patients who were newly prescribed with pirfenidone at the time of participation in the active surveillance.
Period: Overall Study
Arm/Group | All Nintedanib Treated Patients (Group B + Group C) | Group II- Pirfenidone Patients | Group III - Pirfenidone Patients
Started | 14 | 4 | 3
Completed (Completed the study) | 2 | 0 (Patients were not followed after the baseline visit as it was planned in the protocol.) | 0 (Patients were not followed after the baseline visit as it was planned in the protocol.)
Not Completed | 12 | 4 | 3
Not completed — Other than listed | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Patient refusal to continue taking trial medication | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Change to other medication | 2 | 0 | 0
Not completed — Patients were not followed as planned in the protocol | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Entered Set: Includes patients in screened set who met the eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | All Nintedanib Treated Patients (Group B + Group C) | Group II- Pirfenidone Patients | Group III - Pirfenidone Patients | Total
Number analyzed (Participants) | 14 | 4 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (9.59) | 65.3 (4.57) | 68.0 (12.29) | 65.3 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 0 | 6
  Male | 8 | 4 | 3 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of All ADRs in Nintedanib Treated Patients
Description: Incidence of all Adverse Drug Reactions (ADRs) in nintedanib treated patients is reported. An adverse reaction is defined as at least a reasonable possibility of a causal relationship between a suspected medicinal product and an adverse event.
  Incidence rate was calculated using the number of patients with ADRs events per treatment divided by time at risk expressed as [100 patient-years (pt-yrs)].
  Time at risk was calculated as below:
  If patients with AE: Time at risk= (start date of first AE- start date of treatment administration) +1; If patients without AE: Time at risk= (end of date at risk (date of study completion or date of discontinuation or last visit date available)-start date of treatment administration) +1.
Time Frame: From the day Nintedanib was initiated until 52 weeks, up to 52 weeks.
Population: Treated Set: Patients who met all eligibility criteria and have taken at least one dose of nintedanib.
  Outcome measures were not collected for pirfenidone treated patients, since per study protocol for the pirfenidone treated patients only baseline characteristics data were planned to be collected. After the baseline visit the pirfenidone treated patents were not followed.
Measure: Number (95% Confidence Interval); unit: patients with ADR events/100 pt-years
Arm/Group | All Nintedanib Treated Patients (Group B + Group C)
Number analyzed (Participants) | 14
patients with ADR events/100 pt-years | 11.0 [0.28 to 61.46]

2. Primary Outcome: Incidence Rate of All SAEs in Nintedanib Treated Patients
Description: Incidence rate of all Serious Adverse Events (SAEs) in nintedanib treated patients is reported.
  A SAE was defined as any adverse event which:
  * results in death,
  * is life-threatening,
  * requires in-patient hospitalization, or
  * prolongation of existing hospitalisation,
  * results in persistent or significant disability or incapacity, or
  * is a congenital anomaly/birth defect.
  Incidence rate was calculated using the number of patients with SAEs events per treatment divided by time at risk expressed as [100 patient-years (pt-yrs)].
  Time at risk was calculated as below:
  If patients with AE: Time at risk= (start date of first AE- start date of treatment administration) +1; If patients without AE: Time at risk= (end of date at risk (date of study completion or date of discontinuation or last visit date available)-start date of treatment administration) +1.
Time Frame: From the day Nintedanib was initiated until 52 weeks, up to 52 weeks.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: patients with SAEs events/100 pt-years
Arm/Group | All Nintedanib Treated Patients (Group B + Group C)
Number analyzed (Participants) | 14
patients with SAEs events/100 pt-years | 11.4 [0.29 to 63.65]

3. Secondary Outcome: Percentage of Patients With AEs Leading to Permanent Dose Reductions of Study Drug
Description: Percentage of patients with Adverse Events (AEs) leading to permanent dose reductions of study drug is reported.
Time Frame: From the day Nintedanib was initiated until 52 weeks, up to 52 weeks.
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | All Nintedanib Treated Patients (Group B + Group C)
Number analyzed (Participants) | 14
percentage of patients | 0

4. Secondary Outcome: Percentage of Patients With AEs Causing Dose Interruption of Study Drug
Description: Percentage of patients with Adverse Events (AEs) causing dose interruption of study drug is reported.
Time Frame: From the day Nintedanib was initiated until 52 weeks, up to 52 weeks.
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | All Nintedanib Treated Patients (Group B + Group C)
Number analyzed (Participants) | 14
percentage of patients | 0

5. Secondary Outcome: Percentage of Patients With AEs Leading to Permanently Discontinuation of Study Drug
Description: Percentage of patients with adverse events (AEs) leading to permanently discontinuation of study drug is reported.
  Percentages are rounded to one decimal places.
Time Frame: From the day Nintedanib was initiated until 52 weeks, up to 52 weeks.
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | All Nintedanib Treated Patients (Group B + Group C)
Number analyzed (Participants) | 14
percentage of patients | 7.1

ADVERSE EVENTS:
Time Frame: From the day Nintedanib was initiated until 52 weeks, up to 52 weeks.
Description: Treated Set: Patients who met all eligibility criteria and have taken at least one dose of nintedanib. Adverse events were not collected for pirfenidone treated patients, since per study protocol for the pirfenidone treated patients only baseline characteristics data were planned to be collected. After the baseline visit the pirfenidone treated patents were not followed.
Arm/Group | All Nintedanib Treated Patients (Group B + Group C)
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Nintedanib Treated Patients (Group B + Group C) (N=14)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Nintedanib Treated Patients (Group B + Group C) (N=14)
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03047031/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03047031/SAP_001.pdf